CLINICAL TRIAL: NCT04221646
Title: Effect on BTL-899 Device for Non-invasive Lipolysis on Human Thighs and Saddlebags
Brief Title: Non-invasive Lipolysis on Human Thighs and Saddlebags
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTL-899THI
Record Dates: First submitted 2019-12-18; First posted 2020-01-09 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Adipose Tissue Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thighs circumference reduction (Experimental): The subjects will be enrolled and treated once per week. Both legs will be treated consecutively. The therapy will be applied simultaneously.
  Interventions: Device: BTL-899
- Saddlebags fat thickness reduction (Experimental): The subjects will be enrolled and treated once per week. Both legs will be treated consecutively. The therapy will be applied consecutively too.
  Interventions: Device: BTL-899

INTERVENTIONS:
Device: BTL-899 — Treatment with study device.

SUMMARY:
The study is a prospective two-arm, open-label, interventional study with four treatment procedures and two follow-up visits.

DETAILED DESCRIPTION:
This study aims to evaluate the clinical safety and efficacy of the BTL-899 device for non-invasive lipolysis and fat reduction in the thigh and saddlebag area. This is a prospective, open-label, two-arm study; therefore the participants will be assigned to two study groups. Each participant will complete 4 treatment visits and 2 follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 20 to 35 kg/m2.
* Visible excess of adipose tissue at the treatment sites (ARM 1 - thigh area; ARM 2 - saddlebags area).
* Subjects willing and able to abstain from partaking in any treatments other than the study procedure to promote body contouring and/or weight loss during study participation.
* No procedure for fat reduction (including cellulite treatment) in the last six months.
* Subjects willing and able to maintain his/her regular (pre-procedure) diet and exercise regimen without effecting a significant change of weight in either direction during study participation.
* Age between 21 and 70 years.

Exclusion Criteria:

* Electronic implants (such as intrauterine device, cardiac pacemakers, defibrillators, and neurostimulators)
* Cardiovascular diseases
* Vascular diseases (such as chronic venous insufficiency, deep venous thrombosis, varicose veins, etc.)
* Femoral or inguinal hernia
* Disturbance of temperature or pain perception
* Pulmonary insufficiency
* Metal implants
* Drug pumps
* Malignant tumor
* Hemorrhagic conditions
* Septic conditions and empyema
* Acute inflammations
* Systemic or local infection such as osteomyelitis and tuberculosis
* Contagious skin disease
* Elevated body temperature
* Pregnancy
* Breastfeeding
* Injured or otherwise impaired muscles
* Scars, open lesions, and wounds at the treatment area
* Basedow's disease
* Previous liposuction in the treatment area in the last six months
* Unstable weight within the last 6 months (change in weight ± 3%)
* Previous body contouring or cellulite treatments in the thighs area in the last six months
* Any other disease or condition at the investigator's discretion

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-13 (Actual)

PRIMARY OUTCOMES:
Changes in Fat Thickness Measured via Ultrasound | 6 months
  To gather clinical evidence that the BTL-899 device is able to induce non-invasive lipolysis when used on thighs and saddlebags. The fat thickness changes will be measured by means of ultrasound.
Participants' Satisfaction Measured Via Questionnaires | 6 months
  Evaluation of the participants' satisfaction with the therapy via Therapy Satisfaction Questionnaires. Global Aesthetic Improvement Scale (Quality of Life questionnaire) will be used where score "3" means "very much improved" and "-3" is "very much worse".
Evaluation of the Therapy's Safety Measured Via Therapy Comfort Questionnaire | 6 months
  The outcome will further be measured through the occurrence of adverse events or lack thereof. On Numerical Analog Scale (0-10), where 0 represents 'no pain' and 10 represents 'worst possible pain' select the level of pain experienced during the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Aesthe Clinic, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No